CLINICAL TRIAL: NCT02381821
Title: The Measurement of Endometrial Volume and Sub-endometrial Vascularity to Replace the Traditional Endometrial Thickness as Predictors of In-vitro Fertilization Success
Brief Title: Endometrial Volume and Sub-endometrial Vascularity as Predictors of In-vitro Fertilization Success
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Maged, Assistant professor, Cairo University
Other Study IDs: 127
Record Dates: First submitted 2015-03-03; First posted 2015-03-06 (Estimated); Last update posted 2018-01-03 (Actual); Status verified 2018-01

CONDITIONS: Reproductive Techniques, Assisted
Keywords: junctional zone; Implantation; Intracytoplasmic sperm injection
MeSH Terms: conditions — Helping Behavior | interventions — Gonadotropin-Releasing Hormone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- pregnant: women undergoing ICSI who became pregnant
  Interventions: Other: 3 D ultrasound and Doppler examination; Drug: GnRH agonist
- Not pregnant: women undergoing ICSI who fail to achieve pregnancy
  Interventions: Other: 3 D ultrasound and Doppler examination; Drug: GnRH agonist

INTERVENTIONS:
Other: 3 D ultrasound and Doppler examination — Endometrial thickness was measured in the longitudinal plane at the widest anteroposterior diameter with a trans-vaginal 2D ultrasound, and then 3D mode was then activated with power Doppler setting for this study standardized using a frequency at 4-9 MHZ pulse repetition frequency at 0.5KHz gain at-3.0 and wall motion filter at 1. The sub-endometrial region was considered to be within 3 mm of the originally defined myometrial-endometrial contour. The endometrial volume (EV) and 3D power Doppler indices below the endometrium were measured using the automated VOCAL™ for the 3D power Doppler histogram analysis
Drug: GnRH agonist — All women received daily subcutaneous 0.1 mg triptorelin injection started from day 21) of the cycle preceding stimulation. Downregulation of the pituitary gonadotropins was confirmed after 12 days , gonadotropin (Gn) induction was started using Human menopausal gonadotropins for ovarian stimulation. The starting dose was 225 to 300 IU . Ultrasound Folliculometry was done every other day . When two or more follicles reached a minimum mean diameter of 18 mm, triggering of ovulation trigger was done using Human chorionic gonadotropin (hCG) 10,000 IU and ovum pick up was scheduled 36 hours later

SUMMARY:
100 patients aged 21-40 years old, diagnosed as primary or secondary infertility These patients are then assigned to receive ICSI treatment (ovulation induction, . They undergo a 3D vaginal ultrasound before treatment to measure the junctional zone thickness and followed up after treatment to determine the rate of implantation.

Intervention(s) All patients will undergo 3D ultrasound to measure the thickness of the junctional zone at day 21 of the cycle.

DETAILED DESCRIPTION:
100 patients aged 21-40 years old, diagnosed as primary or secondary infertility due to the following causes of infertility; ( Pelvic Inflammatory disease, dysovulation , tubal infertility, unexplained infertility, combined infertility or due to male factor ). These patients are then assigned to receive fertility treatment (ICSI) They undergo a 3D vaginal ultrasound before treatment to measure the junctional zone thickness and followed up after treatment to determine the rate of implantation.

Intervention(s) All patients will undergo 3D ultrasound to measure the thickness of the junctional zone at day 21 of the cycle.

ELIGIBILITY:
Inclusion Criteria:

* A normal transvaginal ultrasound is defined as having no visible intracavitary pathology (e.g. submucous myomas, polyps or septa) and was be performed in the follicular phase of the menstrual cycle. Intramural myomas without impression or deformation of the uterine cavity were incorporated in the definition of a normal ultrasound

Exclusion Criteria:

* Exclusion criteria included Females aged above 40 years old , patients with endometriosis, abnormal endocrine functions as Diabetes mellitus, thyroid disorders and adrenal abnormalities ,general diseases, those with ovarian cysts or have azospermic partners

Ages: 19 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: women with primary or secondary infertility and were scheduled for a first IVF/ICSI treatment cycle due to Pelvic Inflammatory disease, ovulatory dysfunction, tubal infertility, unexplained infertility , combined infertility with normal transvaginal ultrasound.
Sampling Method: Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-12-03 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
pregnancy rate | 14 days after embryo transfer